CLINICAL TRIAL: NCT06252766
Title: The Effect of a Clown Accompanying Children During Blood Collection on Pain and Anxiety: A Randomized Controlled Study
Brief Title: A Clown Accompanying Children During Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Semra Kose, Asisstant Proffessor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NecmettinEUHemSK
Record Dates: First submitted 2024-01-23; First posted 2024-02-12 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Child; Therapeutic Play
Keywords: Blood collection; clown; pain; anxiety; pediatric nursing
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled experimental type study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Trio (Researcher, Child and Parent) The researcher, the child and the parent, who knows the groups and waives all rights to the research, will evaluate the children's pain and anxiety levels during the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Clown) (Experimental): During this process, the clown will continue to distract the children by playing games and blowing foam balloons. During the procedure, the child's pain and anxiety score will be evaluated by both the researcher, the parent, and the child. After the procedure is completed, children will be taken out of the blood collection room and taken to the waiting area in the next room, and after being allowed to rest for 1-2 minutes, surveys will be administered to the children.
  Interventions: Behavioral: Experiment (Clown)
- Control (No Intervention): Blood collection will be routine and surveys will be administered 1-2 minutes after the end of the procedure to determine the level of pain and anxiety during the procedure.

INTERVENTIONS:
Behavioral: Experiment (Clown) — Children included in the intervention group will be accompanied by a clown at the door from the moment they enter the intervention room and The child will be made to sit on the blood collection chair by playing games with them. Meanwhile, the nurse will take blood from the child. lasts for about 2-3 minutes. During this process, the clown is constantly playing games and foam will continue to distract you by blowing up balloons. The child's pain and anxiety score during the procedure the researcher will be evaluated by both the parent and the child. After the procedure is finished, the children will be will be taken out of the room and taken to the waiting area in the next room. Afterwards, the children will be asked how much pain and anxiety they felt during the blood collection procedure. After being allowed to rest for 1-2 minutes a questionnaire form will be applied to the children.
  Arms: Experiment (Clown)

SUMMARY:
Children may be exposed to acute and chronic illnesses during their development and may experience negative emotions and They may be exposed to experiences. For the purpose of diagnosis and treatment in a child admitted to hospital due to illness blood sampling causes pain and anxiety. To reduce pain and anxiety pharmacologic and nonpharmacologic methods are preferred in children. Nonpharmacologic methods supportive, cognitive and physical, although they are more preferred than pharmacological methods in order to classify them as such. Various methods are used within the scope of these classifications, among which The method of distraction is more preferred. This study is based on distraction the effect of the clown, which is one of the methods, on pain and anxiety during blood sampling. to determine the impact of the project. It is planned to be conducted as a randomized controlled study and in this study, 5-12 years old with children between the ages of 18 and 18, and the Pediatric Outpatient Clinic at Necmettin Erbakan University Faculty of Medicine. It was planned to be conducted in the blood collection unit. Minimum number of children to be included in the study The intervention group was planned as 28 and the control group as 28, but due to the possibility of data loss, 15 To collect more data, the number of children to be recruited for both groups is targeted to be 32-33. Children will be randomly assigned to the groups and the assignment to the groups will be based on 'stratification and blocked randomization methods' were planned to be used. Sociodemographic characteristics in data collection form, Wong-Baker Faces Pain Scale (WBFPS), Child Anxiety Scale-Dispositional (CAS-D) scales were planned to be used. Obtaining necessary institutional permissions by the researcher and project advisor It is planned to start the project after it is ensured. Research data were collected through face-to-face interviews with the 'Informed Consent Form'. Family 'Informed Voluntary Consent Form' about the research will be informed. In the intervention group, the blood collection process will be carried out with foamy bubbles accompanied by a clown. by playing with the parents. No treatment was applied to the control group and the parents blood sampling will be performed in the presence of the child. Both groups will be administered the WBFPS and CAS-D scales, will be administered by both the researcher and the parent. The research results to be obtained will be published in international SSCI and/or SCI publishing them as scientific articles in journals, organizing national and international conferences, symposiums and contributing to the literature as a result of being presented in seminars, raising awareness in this field, creating a It is aimed to shed light on future research.

DETAILED DESCRIPTION:
Health is the most important element for the continuation of life. In cases of ineffectiveness in maintaining health, children They apply to a health institution by their parents to receive health care. In this process, as well as parents children are also affected. Children, who are exposed to many acute and chronic diseases during their development, are adversely emotions and experiences. Health to regain health Some physical, cognitive and emotional abnormalities may be observed in the child admitted to the institution. In children whose concrete thinking and ability to establish cause and effect relationships are underdeveloped, hospital concept is a great source of stress. People who perceive the disease as a punishment and perceive the hospital as a foreign the child, who sees the health service as an environment, in order to contribute to the diagnosis-treatment process while benefiting from health services. invasive interventions are widely used. Blood causing tissue damage Painful procedures, such as taking, inserting IV catheters, cause pain, anxiety and fear in the child.

Pain; International Association for the Study of Pain Taxonomy Committee (International Association for the Study of Pain=IASP) defines pain as "pain originating from a specific part of the body, with or without tissue damage, "an unpleasant experience that is influenced by one's past experiences". Today, it is evaluated together with fever, pulse, blood pressure and saturation values. pain is characterized as the 5th vital sign. Evaluation of pain in pediatric patients While it is more difficult than in adults, the assessment depends on the child's perception of pain, gender, age, previous pain experiences, the presence of emotions such as fear, sadness and anger, and the hospital, which is an environment they do not like difficulties are experienced depending on the parents' reaction to the pain. Anxiety; According to the Ministry of Health Anxiety Disorders Clinical Protocol, anxiety is defined as fear, excitement, restlessness, panic, feelings that something bad is going to happen; it is also defined as endocrine responses - physical symptoms with the influence of autonomic stimuli; cognitive symptoms characterized by different thoughts symptoms; behavioral symptoms, which are the expression of emotions and thoughts, are also accompanied. Children blood collection the experience of pain during intravenous procedures such as intravenous procedures, the needle staying inside the body, the blood being drawn thoughts that blood will continuously flow from the area, as a result of uncertainties about this process, due to cognitive development Abstract thinking and perception of threats with high emotions bring the feeling of anxiety to the forefront in the child. Thus, like the concept of hospital, the process of taking blood from the child also causes feelings of anxiety, fear and worry in the child. It also causes pain. Physician order Children who apply to the blood collection unit for diagnosis and treatment may cry, scream and leave the unit during the procedure. tendency to behaviors such as attempting to escape, bending and pulling the extremity to be treated, muscle stiffness.

Nurses, who spend long periods of time with children and are responsible for their care and treatment, are also responsible for pain management. control and should be able to manage pain effectively. Blood collection Many different pharmacologic and nonpharmacologic methods are used for pain control in the procedure. Blood collection Emla Cream, which can be used among pharmacological methods during skin absorption by providing absorption from intact skin. It plays an important role in pain control with its ability to block neural transmission from receptors. However, pharmacologic methods require personnel knowledge and skills, are time consuming and costly. nonpharmacologic methods are less preferred than nonpharmacologic methods. Nonpharmacologic methods are not only a treatment method that reduces pain, but also anxiety and depression, also reduces nausea and vomiting; facilitates restful sleep; makes the patient feel well and increases the desire to participate in their own recovery process. In children nonpharmacological methods are analyzed in three classes: supportive, cognitive/behavioral, physical supportive methods; psychosocial care such as watching videos, reading books, family support for the child, physical methods; touch, skin stimulation, massage, hot and cold applications, cognitive methods are the perceptual - It is based on the sensory-behavioral dimension and includes methods such as relaxation and distraction. Frequently used during the blood collection process attention-getting method that reduces symptoms of anxiety, anxiety, fear and pain, as well as economical, practical application easy and reliable, effective method. Hospital for distraction clowns, watching cartoons, playing video games, using kaleidoscopes and virtual reality (VR) goggles are among the methods that can be used.

Clowns interact with children by playing and providing psychosocial support in any environment. While entertaining children and making them laugh during blood sampling, they may experience pain, anxiety levels. A study that 'An evaluation on reducing children's hospital anxiety: Hospital clown project', hospital clowns contributed positively to children's perception of the hospital. provided by the study. A study that 'Virtualization in Medical Procedures for Pediatric Patients Effects of Reality Use: A Review of the Literature', the investigators analyzed the effects of virtual reality, which is a method of attracting attention. Its use during intravenous procedures has been observed to have positive effects on pain, anxiety.

As a result of the review of the researches, it was concluded that psychosocial psychosocial problems in hospitalization, preoperative care hospital clowns providing support had positive effects on the children and as a result, blood collection The integration of clowns, which are not encountered in the units, into the units and their impact on children will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 5-12,
* Volunteering to participate in the research

Exclusion Criteria:

-Having any physical and mental disability

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Characteristics Form | It will be applied for 1-2 minutes after the blood collection is completed.
  In this section, children's descriptive characteristics (age, gender, mother's education level, father's education level, most the time of the last blood collection, the presence of the parent with the child during the blood collection process) is taking.

SECONDARY OUTCOMES:
Wong-Baker Faces Pain Scale (WBFPS) | It will be applied for 1-2 minutes after the blood collection is completed.
  This scale assessing pain intensity is used in children aged 3-18 years. In this scale, facial expressions are accompanied by numerical A pain score is given according to the values, and the numerical rating of the scale ranges from 0 to 10. Facial expressions ranging from smiling (0 = very happy/no pain) to crying (10 = most painful) It shows the feelings. As the score on the scale increases, the intensity of pain increases, and as the score decreases, the intensity decreases. With the drawing showing the meaning of each of the different numbers on the pain scale, the child tells the nurse about the pain he/she is experiencing. more accurately. This scale is a reliable measurement tool for the Turkish population (Tsao and Zeltzer 2008).

OTHER OUTCOMES:
Child Anxiety Scale-Dispositional (CAS-D) | It will be applied for 1-2 minutes after the blood collection is completed.
  The CAS-D is a thermometer-like scale with a bulb at the bottom and horizontal lines with intervals going upwards. The scale tells children that "All your anxious or angry feelings are at the bulb or bottom of the thermometer. "think about it" is the instruction. "If you are feeling a little bit anxious or nervous, the emotions are a little bit up on the thermometer. can go up. If you are very, very worried or tense, emotions can go all the way to the top. How much on the thermometer put a line showing whether he/she is anxious or irritable". To measure state state anxiety (SAS-D), ask the child to say "this moment", the child is asked to mark what he/she feels. Before filling in the CAS-D, the child's sequencing skills are monitored. He/she is asked They are asked to count up, "Which one is bigger, seven or four?".

CONTACTS AND LOCATIONS:
Overall Officials: Semra KÖSE, PhD,RN, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan Üniversitesi Hemşirelik Fakültesi, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keskin, E. , Buldur, E. & Bal Yılmaz, H. (2021). Virtual Reality in Pain Management in Pediatric Patients Effectiveness of Practices: A Systematic Review . Journal of Current Nursing Research,1(3),96-106 .Retrieved from https://dergipark.org.tr/tr/pub/jcnr/issue/68806/1077642 Kürtüncü, M., & Davas, S. (2020). Nonpharmacologic nonpharmacologic anesthesia during blood sampling in children. the use of methods. Journal of Human Sciences, 17(2), 710-719. doi:10.14687/jhs.v17i2.5785 711 Tsao, Jennie C. I., and Lonnie K. Zeltzer. 2008.